CLINICAL TRIAL: NCT06451315
Title: REGISTRY on the Implementation of Artificial Intelligence in the Automatic Analysis of Vascular Network Segmentation
Acronym: IAVASC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Nurea (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/77
Record Dates: First submitted 2024-05-31; First posted 2024-06-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abdominal Aortic Aneurysm (AAA) treated with EndoVascular Aneurysm Repair (EVAR): Male or female ≥18 years of age with AAA treated with EVAR between ≥50mm or ≥5mm increase in 6 months. The subject is legally competent, has been informed of the nature, the scope, and the relevance of the study and has not manifested an opposition to participate. He is available for set-up and proper implementation of follow-up visits (standard of care) throughout the duration of the registry
  Interventions: Procedure: Analyze CTscans pre-operatively by Nurea System; Procedure: Analyze CTscans pre-operatively by hospital practitioner

INTERVENTIONS:
Procedure: Analyze CTscans pre-operatively by Nurea System — CTscans will be analyzed pre-operatively (6 months before intervention) and post-operatively with an early control scan (up to one-month post-EVAR), compared to a 3, 6 and 12-month control scan by system develop by Nurea
Procedure: Analyze CTscans pre-operatively by hospital practitioner — CTscans will be analyzed pre-operatively (6 months before intervention) and post-operatively with an early control scan (up to one-month post-EVAR), compared to a 3, 6 and 12-month control scan by an hospital practitioner

SUMMARY:
The team hypothesizes that fully automatic analysis of AAA could provide increased performance (decreased duration of segmentation with increased reproducibility and decreased inter and intraobserver variability) to detect aortic aneurysmal sac enlargement (volumes and diameters) and predict the risk of complications during the procedure and during follow-up (MAE, MACE, MALE, Stroke) compared to standard methods of measurement relying on approximate maximum sac diameter.

DETAILED DESCRIPTION:
An abdominal aortic aneurysm (AAA) is an abnormal dilation of the abdominal aortic wall. The most catastrophic consequence of AAA increase evolution is aortic rupture, which still results in high morbidity and mortality. Accurate measurement of AAAs is necessary to predict the risk of rupture during evolution, to take adequate decisions to treat or not the patient as well as detect general and technical risk factors and to follow aneurysm sac behavior after endovascular aortic repair (EVAR).

Despite the widespread use of diameter measurements in clinical trials and its ease of ascertainment in clinical practice for monitoring of AAAs; clinical decision-making regarding the timing of aneurysm repair and even surveillance of sac expansion after EVAR, several studies have concluded that the diameter may not be reliable as a rupture risk criterion and that it should be replaced by more specifics criteria.

Volumetric assessment of the aneurysm is bound to be a better predictor of AAA expansion and risk of rupture. Recently, there has been considerable progress in segmentation software, allowing a semi-automatic calculation of accurate volumes from CTAs. However, despite ample evidence, volumetry has largely remained in the research domain and is still not carried out in most institutions. The major reason is that segmentation methods are time-consuming, they do not allow co-registration of interval studies and they require dedicated software and skilled technicians, which may be difficult to organize.

Innovative software PREAVAorta of Nurea company, using artificial intelligence with deep learning approaches, is able to reconstruct automatically the vascular structures from CT scans. As current solutions only reconstruct the lumen, Nurea's software also segments automatically aneurysms and associated thrombus. With this reconstruction, the software is able to provide diameters (and in particular maximum diameters) but also aneurysmal sac volume. It is the first solution providing automatic AAA volume and comparative evolution during follow-up. In addition, the software provides distances between anatomic points, calcification volume and measurement evolutions between different time points. The software also automatically detects and quantifies calcifications and stenosis on peripheral arteries, which is currently evaluated on the same or independent CT scans for predictive factor analysis, especially with regard to stroke risk for carotid stenosis and accesses, technical difficulties and predictors or MACE (Major Adverse Coronary Event) or MALE (Major Adverse Limb Event) for iliac and femoral arteries.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* AAA treated with EVAR between

  * ≥50mm
  * or ≥5mm increase in 6 months
* The subject is legally competent, has been informed of the nature, the scope, and the relevance of the study and has not manifested an opposition to participate.
* Available for set-up and proper implementation of follow-up visits (standard of care) throughout the duration of the registry

Exclusion Criteria:

* Advancing Alzheimer's disease or socially dependent patient
* Opposition to the use of their data for this research
* Life expectancy supposed to be inferior to 2 years
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient came to the vascular surgery unit for his post-operative follow-up visit who have had surgery for Abdominal Aortic Aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
global volume measure of the aneurysm | 6 months before surgery
  global volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
global volume measure of the aneurysm | Day 3
  global volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
global volume measure of the aneurysm | Month 3
  global volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
global volume measure of the aneurysm | Month 6
  global volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
global volume measure of the aneurysm | Month 12
  global volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.

SECONDARY OUTCOMES:
lumen volume measure of the aneurysm | 6 months before surgery
  lumen volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
lumen volume measure of the aneurysm | Day 3
  lumen volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
lumen volume measure of the aneurysm | Month 3
  lumen volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
lumen volume measure of the aneurysm | Month 6
  lumen volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
lumen volume measure of the aneurysm | Month 12
  lumen volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
thrombus volume measure of the aneurysm | 6 months before surgery
  thrombus volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
thrombus volume measure of the aneurysm | Day 3
  thrombus volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
thrombus volume measure of the aneurysm | Month 3
  thrombus volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
thrombus volume measure of the aneurysm | Month 6
  thrombus volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
thrombus volume measure of the aneurysm | Month 12
  thrombus volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
calcification volume measure of the aneurysm | 6 months before surgery
  calcification volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
calcification volume measure of the aneurysm | Day 3
  calcification volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
calcification volume measure of the aneurysm | Month 3
  calcification volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
calcification volume measure of the aneurysm | Month 6
  calcification volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.
calcification volume measure of the aneurysm | Month 12
  calcification volume measure of the aneurysm by CT-scan. Data are retrospectively collected from the preoperative period (6 months before intervention), during hospitalisation and at systematic follow-up visits at 3, 6 and 12 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Eric DUCASSE, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Chirurgie Vasculaire, Hôpital Pellegrin-tripode, CHU de Bordeaux, Bordeaux, France